CLINICAL TRIAL: NCT02814825
Title: A Multi-Center, Prospective, Single-Arm Study of Patients Undergoing a Two or Three Level ACDF Using ViviGen Cellular Bone Matrix in Conjunction With Cervical Allograft Spacers and DePuy Synthes Spine Anterior Cervical Plate Systems
Brief Title: An ACDF Multi-Center Study Using ViviGen Cellular Bone Matrix
Status: Completed | Type: Observational
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: DSS-2015-01
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Cervical Spondylosis; Degenerative Intervertebral Discs; Herniated Disc
Keywords: ViviGen; ACDF; Cervical
MeSH Terms: conditions — Spondylosis; Intervertebral Disc Degeneration; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ViviGen: Patients undergoing a two or three level ACDF using ViviGen Cellular Bone Matrix in conjunction with cervical allograft spacers and DePuy Synthes anterior cervical plate systems.
  Interventions: Other: ViviGen

INTERVENTIONS:
Other: ViviGen — ViviGen Cellular Bone Matrix is a formulation of cryopreserved viable cortical cancellous bone matrix and demineralized bone. ViviGen is a Human Cells, Tissues, and Cellular and Tissue-based Product (HCT/P) as defined by the U.S. Food and Drug Administration in 21 CFR 127 1.3(d).
  Other Names: ViviGen Cellular Bone Matrix

SUMMARY:
The purpose of this post-market study is to collect data on ViviGen and how its use affects fusion rates in the cervical spine when used as additional grafting material to fill the cervical spacer. The patient population of interest is patients who have already elected to undergo a 2-3 level ACDF surgical procedure using ViviGen, per standard of care.

ELIGIBILITY:
Inclusion Criteria:

Candidates who satisfy ALL of the following inclusion criteria and consent to participate in the study may be considered eligible for enrollment:

1. Diagnosed by the investigator with at least one (1) of the following:

   * Symptomatic cervical spondylosis;
   * Degenerative disc disease (DDD), defined as discogenic pain with degeneration of the disc confirmed by history and imaging studies;
   * Herniated nucleus pulposus (HNP)
2. Subjects who are candidates and have already elected to undergo contiguous two or three-level ACDF surgery between C2-C7 of the cervical spine
3. Skeletally mature adults between 21 and 75 years of age
4. Subjects, who, in the opinion of the Investigator, are able to understand the purpose of the study and are willing to return for all the required post-operative standard of care follow-up visits and have their data collected.

Exclusion Criteria:

Candidates who meet ANY of the following exclusion criteria are not considered eligible for study participation:

1. Posterior instrumentation necessary at same levels being treated
2. Instability associated with major reconstructive surgery for primary tumors or metastatic malignant tumors of the cervical spine
3. Instability associated with cervical spine trauma
4. Acute or chronic systemic or localized spinal infections
5. Previous deep anterior cervical surgeries such as thyroid, carotid, or high thoracic surgery (T5 and above)
6. History of previous cervical fusion surgery at greater than one level
7. Previous pseudoarthrosis at any level of the cervical spine
8. Nursing mothers or women who are pregnant or plan to become pregnant during the time of the study
9. Severe osteoporosis (per the Investigator's diagnosis or per a T-score greater than or equal to 2.5 SD below the mean for a young, healthy adult) that may prevent adequate fixation of screws and thus preclude the use of a cervical plate system
10. Subjects who have a known or suspected allergy to any of the following antibiotics and/or reagents: Gentamicin Sulfate, Meropenem, Vancomycin, Dimethyl Sulfoxide (DMSO), and Human Serum Albumin (HSA)
11. Immune compromised subjects
12. Pre-existing neurological abnormalities other than deficits produced by the spinal fusion (e.g. MS, Parkinson's, CVA, diabetic neuropathy, peripheral neuropathy)
13. Conditions that could preclude the possibility of fusion in the Investigator's opinion (e.g. cancer, kidney dialysis, smoking, uncontrolled diabetes, osteopenia)
14. History of pre-operative dysphagia
15. Symptomatic shoulder pathologies under active treatment
16. Known sensitivity to device materials
17. Subjects who, in the opinion of the Investigator, have any other existing condition that would compromise their participation and follow-up in this clinical study

    Intraoperative exclusion criteria:
18. Intraoperative decision by the surgeon to use implants not compatible or cleared for use with ViviGen
19. Intraoperative decision by the surgeon to use other bone grafts substitutes such as DBM or rhBMP

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients with cervical spondylosis, degenerative disc disease (DDD), or herniated nucleus pulposus (HNP) who are to receive cervical spine surgery with anterior column support at two or three contiguous levels (C2-C7)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Fusion | 12 Months
  An independent radiologist will review films to determine fusion

SECONDARY OUTCOMES:
VAS (Visual Analog Scale) | 12 Months
  Patient neck and arm pain reported on a VAS
NDI (Neck Disability Index) | 12 Months
  Functional success based on results from the NDI
SF-12 | 12 Months
  Quality of life using SF-12 questionnaire
OR (Operating Room) Time | 0 Days
  Length of time to complete the two or three level ACDF (Anterior Cervical Discectomy and Fusion) using ViviGen
Length of Hospital Stay | 12 Months
  Length of time the patient remains in the hospital before being discharged after their two or three level ACDF using ViviGen
Return to Work | 12 Months
  How many patients return to work after having their two or three level ACDF using ViviGen
Adverse Events | 12 Months
  Rate of adverse events (AEs)
Time to Fusion | 12 Months
  Time to fusion as assessed by plain films

IPD SHARING:
Plan to Share IPD: No